CLINICAL TRIAL: NCT04191330
Title: Artificial Intelligence Mobile Health Trial Of A Digital Platform To Optimize Guideline Directed Heart Failure Therapy Using Wearable Sensors
Brief Title: Artificial Intelligence Mobile Health Trial Of A Digital Platform To Optimize GDMT Using Wearable Sensors
Acronym: AIM-POWER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biofourmis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BV-EV-HF-1901
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Control (No Intervention): Subjects in the Control Arm will receive standard of care as normally provided in the clinical center where the study is being conducted.
- Intervention (Experimental): Subjects randomized to the Intervention Arm will be remotely monitored for 90 days using the BiovitalsHF platform to manage initiation and titration of GDMT with and outside of normal or traditional clinical encounters.
  Interventions: Device: BiovitalsHF

INTERVENTIONS:
Device: BiovitalsHF — BiovitalsHFTM is a cloud-based platform that incorporates continuous physiology data from remote vital signs monitoring devices and electronic patient reported outcome (ePRO) monitoring of subjects at-home to support GDMT dose titration for HFrEF patients.
  Arms: Intervention

SUMMARY:
The goal of this real-world, multi-center, randomized, outpatient study is to assess the effectiveness of the Biofourmis cloud based BiovitalsHF platform to recommend optimal titration of Guideline-Directed Medical Therapy (GDMT) for heart failure with reduced ejection fraction (HFrEF) subjects.

DETAILED DESCRIPTION:
Patients with heart failure (HF) remain at high risk for hospitalization and death in part due to underuse of guideline directed medical therapy (GDMT). Digital interventions may facilitate rapid initiation, titration and optimization of GDMT but have not been systematically evaluated in randomized control trials. In the AIM-POWER study, we evaluated the safety and efficacy of a novel software medical application, BiovitalsHF, as a strategy to guide remote optimization of GDMT in patients with HF with reduced ejection fraction (HFrEF).

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible to be included in the study only if all the following criteria apply:

* Written informed consent must be obtained before any assessment is performed
* Age ≥ 22 years at signing of informed consent
* Diagnosis of heart failure with left ventricular ejection fraction ≤ 40%, EF can be assessed by any validated method, but assessment must have occurred within the last year.
* HFrEF patient not on optimal GDMT defined as:

Participant not on optimal GDMT for HFrEF per investigator judgement. This would include patients ranging from no treatments for HFrEF to a patient on multiple GDMTs for HFrEF but with at least 1 medication at 50% or less than target dose.

Exclusion Criteria:

Subjects are excluded from the study if any of the following criteria apply:

Therapy related

* Absolute contraindications to HF GDMT Disease related
* Heart failure hospitalization in the past 28 days.
* Baseline creatinine > 2 mg/dl or potassium level at baseline, ≥5 mEq/L or eGFR <30 mL/min/1.73 m2
* Receiving dialysis at screening
* Baseline systolic blood pressure <100 mmHg
* History of heart transplant or on transplant list
* Current or planned left ventricular assist device Comorbidity or other medical conditions
* Uncontrolled asthma
* Active wheezing on physical exam
* Uncontrolled severe COPD
* Diagnosed with cirrhosis
* Currently being treated for active malignancy and life expectancy is less than one year
* Currently receiving hospice or comfort care Prior or concurrent clinical study experience
* Currently participating or receiving treatment in an investigational device or investigational drug study while participating in this study Other General Exclusions
* Subject unable to independently navigate and operate smartphone applications
* Subject not proficient with written and spoken English or Spanish
* Subject determined likely to be non-compliant by physician/HCP
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (e.g., Clinical Outcome Assessments) to the best of the subject and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition, or disease (with the exception of those outlined above) that, in the opinion of the investigator or Biofourmis medical monitor, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
* Subject has diminished decision making capability

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
• To assess the effectiveness of the Biofourmis cloud-based BiovitalsHF DTx to improve guideline-directed medical therapy (GDMT) adoption in subjects with heart failure with reduced ejection fraction (HFrEF) after 90 days of using the platform | 90 days
  The primary endpoint will be the between-group difference in the change at 90 days, between the intervention and control arm in heart failure optimal therapy score.
  Heart Failure Optimal Therapy Score: A heart failure optimal therapy score was developed (see Table S9 below) based on clinical practice guidelines, including the 2021 Update to the 2017 ACC expert consensus decision pathway for optimization of heart failure treatment {REF}. One point is awarded for initiating evidence-based BB, MRA, or ARNI and two points for up titrating those classes of medications to 50% or higher target dose. Two points are awarded for initiating SGLT2 inhibitor as there is a single approved dose (and no opportunity for dose titration). Finally, if a patient is not on an ARNI, one point is awarded for ACEi/ARB at 50% or higher target dose. Of note, ARNI patients do not receive points for ACEi/ARB. The maximum possible score is 8 points, and the minimum possible score is 0 points.

SECONDARY OUTCOMES:
• To assess the effectiveness of the Biofourmis cloud-based BiovitalsHF DTX to improve the composite clinical outcome by calculating the win ratio between treatment and control arm. | 90 days
  A win ratio [13] will be used to analyze the composite endpoints in the following order of clinical importance:
  * Time to CV death
  * Time to heart failure related hospitalization
  * Improvement in GDMT score
  * Improvement in KCCQ score
  * Reduction on NTproBNP by 30% compared to baseline (TABLE 3)
• To assess the effectiveness of the Biofourmis cloud based BiovitalsHF DTx to help improve GDMT adoption and on clinical outcomes. | 90 days
  • The key secondary endpoint will be the percentage of subjects on target dose of GDMT. Comparisons between the control and intervention arm will be based on the CHAMP-HF registry design [4]. At baseline, day 90, and day 180, subjects will be divided into one of four groups according to prescribed dose of GDMT: subjects not receiving medication, subjects treated with <50% target dose, subjects treated with 50 to <100% target dose, and subjects treated with >100% target dose.
GDMT initiation | 90 days
  • Initiation of evidence-based beta-blocker, ACEi/ARB/ARNI, MRA or SGLT2 inhibitors including proportion of subjects switching from ACEi/ARB to ARNI
Quadruple therapy | 90 days
  • Proportion of subjects on 4 GDMT drug classes
Time to GDMT optimization | 90 days
  • Time taken to achieve 50% target dose between control and intervention arms.
Change in biomarkers | 90 days
  • Change in NT-pro-BNP
Safety outcomes | 90 days
  * Incidence of worsening renal function (i.e., defined as an increase in serum creatinine > 0.5 mg/dl)
  * Incidence of symptomatic postural hypotension (defined as dizziness, lightheadedness, or syncope due to low blood pressure)
  * Objective evidence of hypotension (SBP < 90 mmHg)
  * Incidence of hyperkalemia (i.e., defined K ≥ __5.5 mEq/L)
  * Incidence of angioedema
  * Incidence of severe bradycardia (i.e., defined as an average heart rate < 50 bpm for 12 hours in one day or for 4 contiguous hours)

OTHER OUTCOMES:
Change in quality of life and function | 90 days
  • Change in KCCQ-23

CONTACTS AND LOCATIONS:
Overall Officials: Akshay Desai, MD, Study Chair — Brigham and Womens Hospital; Adam Devore, MD, Principal Investigator — Duke Clinical Research Institute
Locations (14):
- United States (14):
  - Cardiology and Medicine Clinic, Little Rock, Arkansas
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Piedmont Athens Regional Medical Center, Athens, Georgia
  - Baptist Health Louisville Heart Failure Clinic, Louisville, Kentucky
  - Cambridge Medical Trials, Alexandria, Louisiana
  - Medstar Union Memorial Hospital, Baltimore, Maryland
  - St Joseph Mercy, Ypsilanti, Michigan
  - Jackson Heart, Jackson, Mississippi
  - University of Medical Center of Southern Nevada, Las Vegas, Nevada
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Premier Cardiovascular Institute, Dayton, Ohio
  - Providence St Vincent Medical Center, Portland, Oregon
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Austin Heart, San Marcos, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeVore AD, Majmudar M, Etters L, Xie J, Hao C, Lam PH, Hernandez AF, Fonarow GC, Desai AS. Digital Platform to Optimize Guideline-Directed Heart Failure Therapy: Results of the AIM-POWER Trial. Circ Heart Fail. 2025 Dec 3:e013231. doi: 10.1161/CIRCHEARTFAILURE.125.013231. Online ahead of print. PMID 41332416